CLINICAL TRIAL: NCT02254486
Title: A Multicenter Randomized Parallel Group Phase III Study Comparing the Bowel Cleansing Efficacy, Safety and Tolerability of NER1006 (a Low Volume Bowel Cleansing Solution) Versus a Trisulfate Bowel Cleansing Solution Using 2-Day Split-Dosing Regimen in Adults
Brief Title: Multicenter Randomized Parallel Group Phase III Study Comparing the Bowel Cleansing Efficacy, Safety and Tolerability of NER1006 Versus Trisulfate Solution Using 2-Day Split-Dosing Regimen in Adults
Acronym: NOCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NER1006-01/2014 (NOCT); 29672 (Other: Quorum Review IRB)
Record Dates: First submitted 2014-10-01; First posted 2014-10-02 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Colon Cancer; Colorectal Carcinoma; Colon Cleansing
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NER1006, 2-Day Split-Dosing (Experimental): NER1006:2-Day Split-Dosing Regimen (to commence in the evening of the day before the colonoscopy)
  Interventions: Drug: NER1006
- Trisulfate Solution, 2-Day Split-Dosing (Active Comparator): Trisulfate Solution 2-Day Split-Dosing Regimen (to commence in the evening of the day before the colonoscopy)
  Interventions: Drug: Trisulfate solution

INTERVENTIONS:
Drug: NER1006 — The subject will self-administer the first dose of the assigned investigational product in the evening prior to the scheduled colonoscopy and take mandatory additional clear fluid. Subject will take the second dose together with mandatory additional clear fluids on the morning of the colonoscopy.
  Arms: NER1006, 2-Day Split-Dosing
Drug: Trisulfate solution — The subject will self-administer the first dose of the assigned investigational product in the evening prior to the scheduled colonoscopy and take mandatory additional clear fluid. Subject will take the second dose together with mandatory additional clear fluids on the morning of the colonoscopy.
  Arms: Trisulfate Solution, 2-Day Split-Dosing

SUMMARY:
This study evaluates the efficacy, safety and tolerability of NER1006 versus Trisulfate Solution (TS) in adult patients requiring bowel cleansing prior to any procedure that requires a clean bowel, using a 2-Day evening/morning Split-Dosing regimen. Approximately 540 patients will be randomised with the aim of achieving a minimum of 245 patients in each of the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female outpatients and inpatients aged ≥18 to ≤85 years undergoing a screening, surveillance, or diagnostic colonoscopy
* Females of child bearing potential must have a negative pregnancy test at Screening and at Visit 2 and must be practising one of the following methods of birth control and agree to continue with the regimen throughout the study period: Oral, implantable, or injectable contraceptives (for a minimum of three months before study entry) in combination with a condom; Intrauterine device in combination with a condom; Double barrier method (condom* and occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/cream/suppository)
* Willing, able and competent to complete study and comply with instructions.

Exclusion Criteria:

* Patients with past history within last 12 months or current episode of severe constipation (requiring repeated use of laxatives/enema or physical intervention before resolution), known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.
* Patients with ongoing severe acute Inflammatory Bowel Disease (IBD).
* Patients who have had previous significant gastrointestinal surgeries, including colonic resection, sub-total colectomy, abdomino-perineal resection, de-functioning colostomy, Hartmann's procedure and de-functioning ileostomy or other similar surgeries involving structure and function of the small or large colon.
* Regular use of laxatives or colon motility altering drugs in the last month (i.e. more than 2-3 times per week) and/or laxative use within 72 hours prior to administration of the preparation.
* Patients with active intestinal bleeding episodes or with a clinically significant low hemoglobin level <9 g/dL for women and <11 g/dL for men at screening.
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Known phenylketonuria.
* Known hypersensitivity to polyethylene glycols, ascorbic acid and sulfates (not including sulfa-based products) or any other component of the investigational product or comparator.
* Past history within the last 12 months or evidence of any on-going clinically relevant electrocardiogram (ECG) abnormalities (e.g. arrhythmias).
* History of uncontrolled hypertension with systolic blood pressure >170 mmHg and diastolic blood pressure >100 mmHg.
* Patients with cardiac insufficiency NYHA grades III or IV.
* Patients with moderate to severe renal insufficiency (i.e. with GFR, <60 mL/min/1.73m2).
* Patient with serum albumin < 3.4 g/dL.
* Patients with liver disease of grades B and C according to the Child Pugh classification.
* Patients suffering from dehydration at screening as evaluated by the Investigator from physical examination and laboratory investigations.
* Patients with clinically significant electrolyte abnormalities, whether pre-existing or noted at screening, such as hypernatremia, hyponatremia, hyperphosphatemia, hypermagnesemia, hypokalemia, hypocalcaemia, dehydration, or those secondary to the use of diuretics or angiotensin converting enzyme (ACE) inhibitors.
* Patients with any other clinically significant hematological parameters including coagulation profile at screening.
* Patients with impaired consciousness that might predispose them to pulmonary aspiration.
* Patients undergoing colonoscopy for foreign body removal and/or decompression.
* Patients who are pregnant or lactating, or intending to become pregnant during the study.
* Clinically relevant findings on physical examination based on the Investigator's judgment.
* History of drug or alcohol abuse within the 12 months prior to dosing.
* Concurrent participation in an investigational drug or device study or participation within three months of study entry.
* Patients who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures, e.g. cognitively impaired, debilitated or fragile patients.
* Patients who are ordered to live in an institution on court or authority order.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Demicco, Principal Investigator — Anaheim Clinical Trials, CA
Locations (12):
- United States (12):
  - Anaheim Clinical Trials, Anaheim, California
  - Investigative Clinical Research, Annapolis, Maryland
  - MGG Group Co., Inc., Chevy Chase Clinical, Chevy Chase, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Long Island Gastrointestinal Research Group, LLP, Great Neck, New York
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Investigative Clinical Research, LLC, Mentor, Ohio
  - Advanced Research Institute, Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeMicco MP, Clayton LB, Pilot J, Epstein MS; NOCT Study Group. Novel 1 L polyethylene glycol-based bowel preparation NER1006 for overall and right-sided colon cleansing: a randomized controlled phase 3 trial versus trisulfate. Gastrointest Endosc. 2018 Mar;87(3):677-687.e3. doi: 10.1016/j.gie.2017.07.047. Epub 2017 Aug 10. PMID 28803744
- [Derived] Cash BD, Allen C, Poppers DM. Transient alterations in plasma sodium concentrations with NER1006 bowel preparation: an analysis of three phase III, randomized clinical trials. BMC Gastroenterol. 2022 Sep 5;22(1):412. doi: 10.1186/s12876-022-02484-7. PMID 36064325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial recruited out/in-patients at 12 medical centres in the USA, from September 2014 to May 2015.
Groups:
- Trisulfate Solution 2-Day Split-Dosing: Trisulfate solution: Trisulfate solution 2-Day Split-Dosing Regimen (to commence in the evening of the day before the colonoscopy)
- NER1006 2-Day Split-Dosing: NER1006: NER1006 2-Day Split-Dosing Regimen (to commence in the evening of the day before the colonoscopy)
Period: Overall Study
Arm/Group | Trisulfate Solution 2-Day Split-Dosing | NER1006 2-Day Split-Dosing
Started | 311 | 310
Completed | 261 | 255
Not Completed | 50 | 55
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 2 | 4
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 17 | 15
Not completed — GFR<60mL/min | 16 | 21
Not completed — Various | 12 | 12

BASELINE CHARACTERISTICS:
Population: The number of participants for analysis, 245 per arm, was based on assumed overall cleansing success rates of 90% for both Trisulfate Solution (TS) and NER1006, a non-inferiority (NI) margin of 10%, and at least 90% power to demonstrate NI. The overall number of participants analyzed was based on the modified full analysis set (mFAS).
Groups:
- Total: Total of all reporting groups
Arm/Group | Trisulfate Solution 2-Day Split-Dosing | NER1006 2-Day Split-Dosing | Total
Number analyzed (Participants) | 311 | 310 | 621
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 238 | 243 | 481
  >=65 years | 72 | 67 | 139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (10.56) | 57.7 (10.36) | 57.5 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 152 | 294
  Male | 169 | 158 | 327

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Successful Bowel Cleansing (Overall Colon)
Description: The overall quality of bowel cleansing was assessed by a blinded central reader (an experienced and trained colonoscopist) using the segmental scores of the Harefield Cleansing Scale (HCS). A final HCS grading of A, B, C or D was derived. Grades A and B are classified as successful (i.e., all mucosa could be visualised) and C and D are classified as unsuccessful. Comparison of overall success of cleansing with NER1006 versus Trisulfate solution was evaluated using a non-inferiority study design.
Time Frame: Two days (from day of first dosing to day of colonoscopy)
Population: The overall number of participants analyzed was based on the mFAS. This included all randomized patients, except any patient who (i) was randomized but subsequently failed to meet entry criteria and (ii) in whom it was confirmed (from their patient diary) that the same patient did not receive any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Trisulfate Solution 2-Day Split-Dosing | NER1006 2-Day Split-Dosing
Number analyzed (Participants) | 280 | 276
Participants
  Successful | 238 | 235
  Failure | 42 | 41
Statistical Analysis 1: Comparison: Trisulfate Solution 2-Day Split-Dosing vs NER1006 2-Day Split-Dosing; The hypothesis was to demonstrate NI of NER1006 to Trisulfate Solution (TS) (10% margin). Success rate was number of patients with successful overall bowel cleansing as proportion of number of patients in each group. Treatment effect was NER1006 success rate - TS success rate. A Hochberg procedure was used to control Type I error since there were 2 alternative primary endpoints. An alpha level of 1.25% 1-sided was used. A closed testing procedure used to evaluate superiority if NI was met; Test type: Non-Inferiority or Equivalence — The confidence limits were adjusted for multiple comparisons (two alternative primary endpoints): To be declared non-inferior, the primary endpoint must show a difference in success rates of no greater than 10% in favor of Trisulfate Solution using lower 1-sided 97.5% confidence limits. Calculated using exact Clopper-Pearson confidence limits; p = 0.528, Fisher Exact — P-value adjusted for multiple comparisons (two alternative primary endpoints): To be declared superior, the primary endpoint must demonstrate non-inferiority with 1-sided p-value <0.025, the threshold for statistical significance; Difference in success rate = 0.14, 97.5% CI 1-sided [lower limit -8.15]

2. Primary Outcome: Number of Patients With 'Excellent Plus Good' (Highly Effective) Bowel Cleansing (Colon Ascendens)
Description: The overall quality of bowel cleansing was assessed by a blinded central reader (an experienced and trained colonoscopist) using the segmental scores of the Harefield Cleansing Scale (HCS). Highly effective cleansing in the colon ascendens corresponded to scores 3 (Good) or 4 (Excellent) of the HCS. Adequate plus failure of cleansing corresponded to score 0-2. Comparison of 'Excellent plus good' cleansing of the colon ascendens using NER1006 versus Trisulfate Solution was evaluated using a non-inferiority study design.
Time Frame: Two days (from day of first dosing to day of colonoscopy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Trisulfate Solution 2-Day Split-Dosing | NER1006 2-Day Split-Dosing
Number analyzed (Participants) | 280 | 276
Participants
  Excellent plus good | 82 | 99
  Adequate plus failure | 198 | 177
Statistical Analysis 1: Comparison: Trisulfate Solution 2-Day Split-Dosing vs NER1006 2-Day Split-Dosing; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The confidence limits were adjusted for multiple comparisons (two alternative primary endpoints): To be declared non-inferior the primary endpoint must show a difference in success rates of no greater than 10% in favour of Trisulfate Solution using lower 1-sided 97.5% confidence limits. Calculated using exact Clopper-Pearson confidence limits; p = 0.059, Fisher Exact — P-value was adjusted for multiple comparisons (two alternative primary endpoints): To be declared superior, primary endpoint must demonstrate non-inferiority and with 1-sided p-value <0.025; the threshold for statistical significance; Difference in excellent plus good rate = 6.58, 97.5% CI 1-sided [lower limit -1.69]

3. Secondary Outcome: Adenoma Detection Rate (Colon Ascendens)
Description: Comparison of the number of patients with at least one adenoma detected in the colon ascendens when NER1006 is used for bowel cleansing versus Trisulfate Solution. Adenoma detection rate (ADR) defined as the number of patients with at least one adenoma in the colon ascendens.
Time Frame: Two days (from day of first dosing to day of colonoscopy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Trisulfate Solution 2-Day Split-Dosing | NER1006 2-Day Split-Dosing
Number analyzed (Participants) | 280 | 276
Participants
  Patients with no adenomas detected | 232 | 237
  Patients with at least one adenoma detected | 48 | 39
Statistical Analysis 1: Comparison: Trisulfate Solution 2-Day Split-Dosing vs NER1006 2-Day Split-Dosing; If at least one of the alternative primary endpoints was met, then key secondary endpoints for the same colon region as met by the primary endpoint were evaluated hierarchically in a pre-specified order. The difference in ADR was calculated as NER1006 rate - TS rate using 1-sided 97.5% confidence limits. Formal testing was to proceed in the hierarchy if preceding key secondary endpoint met non-inferiority. This procedure ensured overall Type I error control at 2.5% 1-sided; Test type: Non-Inferiority or Equivalence — To be declared non-inferior, the key secondary endpoint must show a difference in rates of no greater than 10% in favor of Trisulfate Solution using lower 1-sided 97.5% confidence limits. Calculated using exact Clopper-Pearson confidence limits; p = 0.863, Fisher Exact — To be declared superior, the key secondary endpoint must demonstrate non-inferiority and show a significant advantage for NER1006 relative to Trisulfate Solution with 1-sided p-value <0.025, the threshold for statistical significance; Difference in ADR = -3.01, 95% CI 2-sided [-11.36 to 5.28]

4. Secondary Outcome: Adenoma Detection Rate (Overall Colon)
Description: Comparison of the number of patients with at least one adenoma detected in the overall colon when NER1006 is used for bowel cleansing versus Trisulfate Solution. ADR defined as the number of patients with at least one adenoma in the overall colon.
Time Frame: Two days (from day of first dosing to day of colonoscopy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Trisulfate Solution 2-Day Split-Dosing | NER1006 2-Day Split-Dosing
Number analyzed (Participants) | 280 | 276
Participants
  Patients with no adenomas detected | 182 | 183
  Patients with at least one adenoma detected | 98 | 93
Statistical Analysis 1: Comparison: Trisulfate Solution 2-Day Split-Dosing vs NER1006 2-Day Split-Dosing; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.660, Fisher Exact — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Polyp Detection Rate (Colon Ascendens)
Description: Comparison of the number of patients with at least one polyp detected in the colon ascendens when NER1006 is used for bowel cleansing versus Trisulfate Solution. Polyp detection rate (PDR) defined as the number of patients with at least one polyp in the colon ascendens.
Time Frame: Two days (from day of first dosing to day of colonoscopy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Trisulfate Solution 2-Day Split-Dosing | NER1006 2-Day Split-Dosing
Number analyzed (Participants) | 280 | 276
Participants
  Patients with no polyps detected | 213 | 225
  Patients with at least one polyp detected | 67 | 51
Statistical Analysis 1: Comparison: Trisulfate Solution 2-Day Split-Dosing vs NER1006 2-Day Split-Dosing; If at least one of the alternative primary endpoints was met, then key secondary endpoints for the same colon region as met by the primary endpoint were evaluated hierarchically in a pre-specified order. The difference in PDR was calculated as NER1006 rate - Trisulfate Solution rate using 1-sided 97.5% confidence limits. Formal testing was to proceed in the hierarchy if preceding key secondary endpoint met non-inferiority. This procedure ensured overall Type I error control at 2.5% 1-sided; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.953, Fisher Exact — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: Polyp Detection Rate (Overall Colon)
Description: Comparison of the number of patients with at least one polyp detected in the overall colon when NER1006 is used for bowel cleansing versus Trisulfate Solution. PDR defined as the number of patients with at least one polyp in the overall colon.
Time Frame: Two days (from day of first dosing to day of colonoscopy)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Trisulfate Solution 2-Day Split-Dosing | NER1006 2-Day Split-Dosing
Number analyzed (Participants) | 280 | 276
Participants
  Patients with no polyps detected | 144 | 150
  Patients with at least one polyp detected | 136 | 126
Statistical Analysis 1: Comparison: Trisulfate Solution 2-Day Split-Dosing vs NER1006 2-Day Split-Dosing; If at least one of the alternative primary endpoints were met, then key secondary endpoints were evaluated hierarchichally in a pre-specified order. Non-inferiority was concluded if the 1-sided 97.5% confidence limit (CL) for difference in proportion of events between 2 groups excluded a 10% or greater difference was in favor of Trisulate Solution. Formal testing was to proceed in the hierarchy if preceding key secondary endpoint had at least met non-inferiority; Test type: Non-Inferiority or Equivalence — Formal hierarchical testing of this key secondary endpoints was not performed due to the results of the non-inferiority analysis; p = 0.781, Fisher Exact

ADVERSE EVENTS:
Time Frame: Afternoon of Day 1 (first dose) to Day 9 (final clinic visit)
Description: Safety analyses were based on the safety population which included all randomized patients for whom it could not be ruled out (from their patient diary) that they received study drug at least once (n=527). The analyses are based on treatment emergent adverse events (TEAEs). There were no deaths and neither of the serious TEAEs was related to treatment.
Arm/Group | Trisulfate Solution 2-Day Split-Dosing | NER1006 2-Day Split-Dosing
All-Cause Mortality (participants affected / at risk) | 0/265 | 0/262
Serious Adverse Events (participants affected / at risk) | 1/265 | 1/262
Other Adverse Events (participants affected / at risk) | 32/265 | 73/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trisulfate Solution 2-Day Split-Dosing (N=265) | NER1006 2-Day Split-Dosing (N=262)
Gastrintestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trisulfate Solution 2-Day Split-Dosing (N=265) | NER1006 2-Day Split-Dosing (N=262)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal Tenderness (Gastrointestinal disorders) | 1 (1) | 6 (7)
Gastritis (Gastrointestinal disorders) | 3 (3) | 3 (3)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (6) | 18 (19)
Vomiting (Gastrointestinal disorders) | 7 (8) | 16 (16)
Glomerular filtration rate decreased (Investigations) | 5 (5) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 8 (8)
Headache (Nervous system disorders) | 2 (2) | 5 (5)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Fatigue (General disorders) | 3 (3) | 4 (4)

LIMITATIONS AND CAVEATS:
Imputation of failure occurred in 7% of patients. This strict analytical approach reduced the cleansing success rates for both treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No